CLINICAL TRIAL: NCT00606931
Title: Pilot Clinical Study to Evaluate High Resolution PET Imaging- Guidance for Sampling of Breast Abnormalities in Patients With Known or Suspected Breast Cancer
Brief Title: Pilot Study to Evaluate High Resolution PET Image-Guidance for Sampling of Breast Abnormalities
Acronym: PEM-BX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naviscan PET Systems (Industry)
Collaborators: American Radiology Services, Inc (Other); Boca Raton community Hospital, FL (Unknown); Diversified Specialty Institutes, Bensalem, PA (Unknown); Advanced Breast Care Imaging (Industry); Epic Imaging (Industry)
Responsible Party: Judith Kalinyak, MD. Ph.D, Medical Director, Naviscan PET Systems, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEM-07-02; NIH/NCI 5 R44 CA082042-03
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer
Keywords: biopsy; PET; image-guidance; breast cancer; FDG; PEM
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm (Experimental)
  Interventions: Device: Stereo Navigator Accessory to PEM Flex PET Scanner

INTERVENTIONS:
Device: Stereo Navigator Accessory to PEM Flex PET Scanner — For patients with suspicious breast abnormalities seen on high resolution PET image, the patients will be biopsied using commercial vacuum biopsy devices (pre-validated to work with Stereo Navigator) using Naviscan's Stereo Navigator (interventional device) for PET image guidance.

SUMMARY:
The purpose of this pilot clinical study is to test a methodology for using high-resolution Positron Emission Tomography (PET) imaging to guide vacuum-assisted core biopsy of breast abnormalities identified on PET. In order to implement the PET guidance, the study uses the Stereo Navigator accessory to the high-resolution organ-specific PET scanner (PEM Flex™ PET Scanner, Naviscan PET Systems, Inc., San Diego, CA). The Stereo Navigator is an investigational device intended for guiding biopsy needles toward lesions in breasts identified by a physician on a high resolution PET image. The study will evaluate the clinical utility of the Stereo Navigator in guiding the vacuum-assisted core biopsy of breast abnormalities, following the example of prior studies of breast biopsy guided by magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
The study will invite participation from human subjects with newly diagnosed or suspected breast cancer who have one or more breast abnormalities moderately suspicious or highly suggestive of malignancy on breast imaging and requiring biopsy (the lesion(s) of interest). Prospective subjects will be asked to sign IRB-approved consent forms, explaining the use of PET imaging for guiding biopsy of suspicious lesion(s). Up to 30 patients will be recruited in the study. The study will be terminated after approximately 20 subjects undergo PET-guided interventional procedures. In the course of the study, a subject will be injected with 18F-FDG and imaged using the PEM Flex PET scanner. Once an abnormality requiring biopsy is identified on the PET scan, the physician conducting the procedure will use the PET image to plan the biopsy trajectory using the Stereo Navigator Software Module, and use the Stereo Navigator Needle Guide Holder to guide insertion of the introducing stylet toward the lesion. The sampling will be performed using commercially available core biopsy tools routinely used for MRI-guided biopsy.Immediately after the PET-guided biopsy, conventional biopsy markers will be inserted at the biopsy site(s) for correlation with other imaging modalities. Placement of the biopsy marker will be documented using mammography, as per standard clinical practice. Histopathologic results will be correlated with imaging findings. The procedure may be repeated for additional lesions identified on PET at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 25 years or older

* Individuals who have at least one breast imaging finding requiring biopsy, specifically:

  * Individuals who have a breast abnormality(ies) moderately suspicious for or highly suggestive of malignancy on imaging with mammography, ultrasound, or MRI (as per ACR BIRADS™ 4C or 5) and requiring biopsy confirmation OR o Individuals with known breast cancer who have additional imaging abnormality(ies) suspicious for malignancy detected on a high-resolution FDG PET scan
  * Individuals who had recent conventional imaging work-up including x-ray mammography of the breast containing the abnormality of interest.
* Individuals with suspected tumor size measuring one cm or less on mammography and/or ultrasound and/or MRI if the lesion is visible on any of these modalities, except that each site may enroll up to three patients each where the lesion of interest as measured on mammography (or ultrasound and/or MRI if not detectable on mammography) is more than 1 cm. (Note: The study will target patient enrollment such that at least 50% of the lesions to undergo biopsy across all sites will be less than 1 cm in diameter as measured on mammography, or as measured by other modalities, such as ultrasound, CT, or MRI, if the lesion is not detectable or measurable on mammography.)
* Individuals who have agreed to participate in the study and who have signed study-specific informed consent

Exclusion Criteria:

* Women who are or may be pregnant
* Women who are currently lactating or discontinued breastfeeding < 2 months prior to the study
* Age less than 25 years
* Individuals with breast implant(s) in the breast containing the lesion of interest
* Individuals who are scheduled for a sentinel node procedure using radioactive Tc-99m within 24 hours of PET-guided biopsy
* Patients with contraindications for core biopsy and other invasive procedures such as blood coagulation disorders, infection, or who are unwilling to discontinue use of anticoagulant medication prior to the procedure
* Individuals with Type I or poorly controlled Type II diabetes mellitus
* Individuals with a blood glucose level that is above 140 mg/dl at the time of PEM imaging
* Inability to provide informed consent
* Individuals who have had surgery on the study breast(s) within the past 12 months

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E Kalinyak, MD, Ph.D, Principal Investigator — Naviscan PET Systems, Inc
Locations (5):
- United States (5):
  - Boca Raton Community Hospital, Boca Raton, Florida
  - American Radiology Services, Greenspring, Timonium, Maryland
  - Epic Imaging, Portland, Oregon
  - Advanced Breast Care Imaging, Allentown, Pennsylvania
  - Diversified Specialty Institutes, Bensalem, Pennsylvania

REFERENCES:
- [Derived] Kalinyak JE, Schilling K, Berg WA, Narayanan D, Mayberry JP, Rai R, Dupree EB, Shusterman DK, Gittleman MA, Luo W, Matthews CG. PET-guided breast biopsy. Breast J. 2011 Mar-Apr;17(2):143-51. doi: 10.1111/j.1524-4741.2010.01044.x. Epub 2011 Jan 31. PMID 21276128
- See also: Website of Study sponsor : Naviscan PET Systems, Inc — http://www.naviscanpet.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between January & July 2008 at the medical center where they underwent PEM imaging.
Pre-assignment Details: The first enrolled participant was excluded from the analysis, the subject signed the consent form prior to the trial being officially released.
Groups:
- PET Guided Biopsy: No comparison group. All enrolled participants were expected to undergo PET guided biopsy.
Period: Overall Study
Arm/Group | PET Guided Biopsy
Started | 22
Completed | 19
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | PET Guided Biopsy
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions That Were Successfully Biopsied Using the PET-guided Biopsy Method.
Description: Success in completion of the PET guided biopsy of a suspicious lesion was determined by
  1. Alteration in lesion morphology (no change in vs change in lesion morphology) after sampling AND/OR
  2. Visualization of regions with high radioactive uptake within the biopsy specimen consistent with target lesion (focal uptake present vs absent).
Time Frame: within two days of obtaining histopathology of the lesion biopsied
Population: All participants who completed the PET-guided biopsy for a suspicious lesions. 24 lesions were biopsied in 19 participants
Measure: Number; unit: Number of lesions
Arm/Group | PET Guided Biopsy
Number analyzed (Participants) | 19
Number of lesions | 24

2. Secondary Outcome: Number of Participants Who Reported Serious Adverse Events After the PET-Guided Biopsy
Description: Serious Adverse Events are defined as events that
  * Are fatal or life-threatening
  * Require in-patient hospitalization or prolong hospitalization
  * Result in permanent or significant disability/incapacity
  * Result in congenital abnormality/birth defect
Time Frame: Within one week of completing PET-guided biopsy
Measure: Number; unit: Participants
Arm/Group | PET Guided Biopsy
Number analyzed (Participants) | 19
Participants | 0

3. Other Pre Specified Outcome: Number of Participants Who Tolerated the PET-Guided Biopsy Procedure
Description: Participants who could tolerate the procedure and complete it. This was ascertained by patient feedback questionnaire asking for overall discomfort rating from 0 to 5, where 0 is no discomfort and 5 was assigned to acute discomfort that prevented subject from completing the procedure.
Time Frame: Within one week of completing PET-guided biopsy
Measure: Number; unit: Participants
Arm/Group | PET Guided Biopsy
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Arm/Group | PET Guided Biopsy
Serious Adverse Events (participants affected / at risk) | 0
Other Adverse Events (participants affected / at risk) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | PET Guided Biopsy
Nausea (Investigations) | 1/19 (1)
Bruising (Injury, poisoning and procedural complications) | 1/19 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results pending FDA approval or clearance.